CLINICAL TRIAL: NCT00893997
Title: Phase 2 Study of Proteinase 3 PR1 Peptide Vaccine in Myelodysplastic Syndrome (MDS)
Brief Title: PR1 Vaccination in Myelodysplastic Syndrome (MDS)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The trial was ended per sponsor due to slow accrual rates.
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: The Vaccine Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2005-0913
Record Dates: First submitted 2009-05-04; First posted 2009-05-06 (Estimated); Results first posted 2011-04-12 (Estimated); Last update posted 2012-07-16 (Estimated); Status verified 2012-07

CONDITIONS: Leukemia; Myelodysplastic Syndrome
Keywords: myelodysplastic syndrome; MDS; PR1 Peptide Vaccine
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PR-1 vaccine (Experimental): 4 injections of 0.5 mg PR1 peptide vaccine every 3 weeks.
  Interventions: Biological: PR-1 vaccine

INTERVENTIONS:
Biological: PR-1 vaccine — 0.5 mg injections under the skin once every 3 weeks for a total of 4 vaccinations.
  Other Names: PR1 Peptide Vaccine

SUMMARY:
Primary aim:

1. To determine the immunologic response, using a PR1-HLA-A2 tetramer assay, to 4 subcutaneous (SQ) injections of TVC-PR1 vaccine formulated in Montanide ISA 51 VG followed by granulocyte macrophage colony-stimulating factor (GM-CSF) in low risk and intermediate-1 myelodysplastic syndrome (MDS) patients.

Secondary aims:

1. To determine if non-immunologic responders to 4 subcutaneous (SQ) injections of TVCPR1 vaccine formulated in Montanide ISA 51 VG followed by GM-CSF can be converted to immunologic responders by administering 4 additional doses of TVC-PR1 vaccine formulated in Montanide ISA 51 VG followed by GM-CSF.
2. To determine the clinical response to 4 or 8 subcutaneous (SQ) injections of TVC-PR1 vaccine formulated in Montanide ISA 51 VG followed by GM-CSF in patients low risk and intermediate-1 MDS.

DETAILED DESCRIPTION:
MDS cells over-produce proteins found in normal bone marrow cells. These proteins can be used to stimulate the body's immune system to kill the MDS cells. PR-1 is a peptide derived from a protein, and PR1 peptide vaccine is given to help immune cells kill MDS cells. The vaccine is given together with granulocyte macrophage colony stimulating factor (GM-CSF), which increases production of white blood cells and is intended to increase the number of immune cells.

Before you can start treatment on the study, you will have "screening tests." These tests will help the doctor decide if you are eligible to take part in the study. You will have a bone marrow aspirate (about 1 tablespoon) for routine tests and for special studies. To collect a bone marrow aspirate, an area of the hip is numbed with anesthetic and a small amount of bone marrow is withdrawn through a large needle. Blood (about 6 tablespoons) will be drawn. The blood tests are being done to compare pre-treatment blood counts to post-treatment counts, and the aspirate is being done to allow comparison of the number of MDS cells before and after treatment. Both the blood counts and aspirate will show whether the therapy was successful. Women who are able to have children must have a negative blood pregnancy test.

If you are found to be eligible to take part in this study, you will receive the PR-1 vaccine as an injection under the skin once every 3 weeks. You will receive a total of 4 vaccinations. Each vaccination requires 4 shots: 2 of PR-1 vaccine and 2 of GM-CSF. GM-CSF is given to increase the number of immune cells that might respond to the vaccine and eventually kill MDS cells. PR-1 vaccine is mixed with montanide ISA 51, which is used to dissolve and stabilize the vaccine.

Blood (about 1 tablespoon) will be drawn for routine tests 1 time every 3 weeks and (about 3 tablespoons) will be drawn each time before you receive the vaccinations and at follow up visits for the length of the study. You will have a bone marrow aspiration 4 weeks after the 4th and 8th vaccinations (about 1 tablespoon) for routine and for the special tests. These tests will allow researchers to find out if the number of immune cells has increased, whether these cells are able to attack the MDS cells, and whether the cells are related to a change in blood counts. At this time (13 weeks from the first PR-1 vaccine), if your immune system is reacting to the vaccinations, no further vaccinations will be given. This is to avoid production of immune cells that might block the effects of the cells already produced by the first 4 vaccinations. If, at this time (13 weeks from the first PR-1 vaccine), your immune system is not reacting to the drug, you will be offered an additional 4 vaccinations. These additional vaccinations will again be given once every 3 weeks. During this time, blood (about 4 tablespoons) will again be drawn once every 3 weeks for routine and special testing.

You will be taken off study at any time if the disease gets worse or intolerable side effects occur.

Twenty-nine (29) weeks after beginning the study, blood (about 1 teaspoon) will be drawn to check for a response to the vaccine. If you have not responded, you will be taken off study.

If you have responded, you will continue to be followed. Follow-up will involve monthly routine blood tests (1 tablespoon of blood) for 6 months. These can be done at home with results sent to M. D. Anderson. Every 3 months, you will return to M. D. Anderson for a bone marrow aspirate and routine blood tests including the special testing studies.

This is an investigational study. This vaccine is authorized for use in research only and is not commercially available. About 30 patients will take part in this multicenter study. About 20 patients will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Must understand and voluntarily sign an informed consent form
2. Age >/= 18 years at the time of signing the informed consent form
3. Must be able to adhere to the study visit schedule and other protocol requirements
4. HLA-A2 positive at one allele
5. Diagnosis of myelodysplastic syndrome (MDS) and must meet all the following criteria
6. French-American-British (FAB) Class Refractory anemia (RA), Refractory Anemia with Excess Blasts (RAEB), refractory anemia with ringed sideroblasts (RARS)
7. World Health Organization(WHO) Classification refractory anemia (RA), refractory anemia with ringed sideroblasts(RARS), refractory cytopenia with multilineage dysplasia (RCMD), refractory cytopenia with ringed sideroblasts (RCMD-RS) , refractory anemia with excess blasts type 1 (RAEB-1)
8. Less than 20% blasts on marrow aspirate
9. International Prognostic Scoring System (IPSS) risk groups Intermediate 1 or transfusion dependent low risk.
10. Both de novo and therapy related MDS are eligible
11. Eastern Cooperative Oncology Group (ECOG) performance status = 0 or 1
12. Women of childbearing potential must have a negative serum pregnancy test within 30 days of starting study drug. A woman of child-bearing potential is a sexually mature woman who has not undergone a hysterectomy or who has not been naturally postmenopausal for at least 24 consecutive months (i.e., who has had menses at any time in the preceding 24 consecutive months)
13. Male or female of child-bearing potential must agree to use adequate contraceptive methods
14. Serum bilirubin < 2 mg/ml
15. Serum creatinine </= 1.5 mg/ml
16. Serum ALT < 2 x upper normal limit
17. anti-neutrophil cytoplasmic antibody (cANCA) negative
18. Not received specific therapy for MDS for 4 weeks. However, supportive therapy is permitted.

Exclusion Criteria:

1. Marrow blasts on aspirate >/= 20%
2. Blood blasts > 1%
3. Inaspirable bone marrow
4. Myelosclerosis occupying >30% of marrow space
5. Iron absence on marrow examination or transferrin saturation <20% and serum ferritin <50ng/ml
6. B-12 deficiency
7. Folate deficiency
8. History of immune related hematological disorder [i.e.,immune thrombopenia purpura(ITP),autoimmune hemolytic anemia ( AIHA)]
9. Other causes of cytopenia not related to MDS (i.e., GI blood loss)
10. Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form or that will place the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret the data
11. Prior allogeneic or syngeneic transplant
12. Prior solid organ transplant
13. Life expectancy severely limited by diseases other than MDS
14. Pregnant or lactating females
15. Prior vaccine therapy for MDS
16. Chronic use (>2 weeks) of greater than physiologic doses of a corticosteroid agent (dose equivalent to >10 mg/day of prednisone) within 30 days of the first day of study drug treatment. (Topical and inhaled corticosteroids are permitted)
17. Prior history of malignancy other than MDS (except basal cell or squamous cell carcinoma or carcinoma in situ of the cervix or breast) unless the subject has been free of disease for >/= 5 years
18. Known allergy to incomplete Freund's adjuvant
19. Experimental therapy, cyclosporine, antithymocyte globulin, or FK506 within 3 months of study entry
20. Treatment with androgenic hormones, danazol, colony stimulating factors, erythropoietin, thalidomide, arsenic trioxide or other agents used to treat MDS within four weeks of the first day of study treatment
21. refractory anemia with excess blasts in transformation (RAEB-t) (French-American British (FAB) criteria ) or refractory anemia with excess blasts type2 (RAEB-2) (World Health Organization (WHO) criteria)
22. Chloroma
23. Hypercalcemia
24. Progressive viral or bacterial infection. Patients are not eligible unless all infections are resolved and the patient has remained afebrile for seven days without antibiotics
25. Cardiac disease of symptomatic nature or cardiac ejection fraction < 40%
26. Symptomatic pulmonary disease or FEV1, FVC and Carbon Monoxide Diffusing Capacity (DLCO) </= 50% predicted
27. History of Wegener's Granulomatosis or vasculitis
28. History of HIV positivity or AIDS
29. Prior history of AML

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2006-07; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Garcia-Manero, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- U.T. M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: 01/09/07 through 03/24/08. All participants recruited at UT MD Anderson Cancer Center.
Pre-assignment Details: Twelve patients were registered, two patients did not receive drug and were not included in the study group therefore ten patients were evaluable.
Period: Overall Study
Arm/Group | PR-1 Vaccine
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | PR-1 Vaccine
Number analyzed (Participants) | 10
Age Continuous [Median (Full Range); unit: years] | 64 [46 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Patient Immunologic Response
Description: Patients assessed after 4th vaccination for immunologic response categorized as 'Immunologic-Responders' or 'Non-Responders.' Immune response defined as an increase of ≥ 0.5 PR1-HLA-A2 tetramer cells/μl compared to the pre study absolute PR1-HLA-A2 tetramer cells/μl. Time period 29 weeks after study entry, with week 0 corresponding to 1st injection, and 8th injection thus being given at week 25, 29 weeks corresponds to 13 weeks after receipt of a 4th injection.
Time Frame: 29 weeks
Population: Analysis on patients treated; study terminated early.
Measure: Number; unit: participants
Arm/Group | PR-1 Vaccine
Number analyzed (Participants) | 10
participants
  Immunological Response | 3
  No Immunological Response | 7

2. Primary Outcome: Number of Patients With Clinical Response
Description: Clinical response based on the International Working Group (IWG) Response Criteria in myelodysplastic syndromes (MDS): 'Complete Response' or Hematologic Improvement' and 'No Clinical Response'. Clinical responses as assessed by standard criteria with bone marrow biopsy, cytogenetic studies (standard chromosome banding) and molecular studies 3 weeks after the last vaccination.
Time Frame: At 29 weeks
Population: Analysis on patients treated; study terminated early.
Measure: Number; unit: participants
Arm/Group | PR-1 Vaccine
Number analyzed (Participants) | 10
participants
  Complete Response | 0
  Hematological Improvement | 1
  No Clinical Response | 9

ADVERSE EVENTS:
Time Frame: 1 year and 11 months
Arm/Group | PR-1 Vaccine
Serious Adverse Events (participants affected / at risk) | 1/10
Other Adverse Events (participants affected / at risk) | 6/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PR-1 Vaccine (N=10)
Allergic Reaction (General disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PR-1 Vaccine (N=10)
Injection site reaction (General disorders) | 4 (5)
Allergic reaction (General disorders) | 1 (1)
Fatigue (General disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Bone pain (General disorders) | 2 (2)
Chill (General disorders) | 1 (1)
Puritis (Skin and subcutaneous tissue disorders) | 1 (1)
Mucositis (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No